CLINICAL TRIAL: NCT07210983
Title: Low-Intensity Pulsed Ultrasound as an Adjunctive Therapy for Bone Regeneration Following Jaw Cyst Enucleation With Curettage: A Randomized Controlled Trial
Brief Title: Low-Intensity Pulsed Ultrasound as an Adjunctive Therapy for Bone Regeneration Following Jaw Cyst Enucleation
Acronym: LIPUS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sadam Elayah (Other)
Collaborators: Sichuan University (Other)
Responsible Party: Sponsor-Investigator, Sadam Elayah, Dr, Sichuan University
Organization: Sichuan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WCHSIRB-D-2021-280-R1; 31570950 (Other Grant/Funding Number: National Nature Science Foundation of China); 2024YFFK0376 (Other Grant/Funding Number: Science and Technology Foundation of Sichuan Province)
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Jaw Cysts; Curettage
Keywords: Bone Regeneration; Hounsfield unit; Jaw Cysts; Low-intensity pulsed ultrasound; Three-Dimensional Volumetric Analysis; Bone Density
MeSH Terms: conditions — Jaw Cysts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Before the group's assignment, all enucleation procedures will be carried out by the same surgeon to ensure consistency in surgical techniques. Three days after the surgery, patients will be randomly allocated to one of two groups using opaque, sealed envelopes. A nurse who is uninvolved in the research will open the randomization envelopes to reveal the assigned treatments: those in the ultrasound group will receive active LIPUS therapy, whereas the control group will be given sham LIPUS therapy, using an inactive device. Throughout the study, the surgeon, participants, outcome assessors, and statistician will remain unaware of the group allocation, maintaining a triple-blind design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound Therapy Will Enhance Bone Healing and Recovery After Jaw Cyst Surgery (Experimental): Ultrasound Therapy Arm (Intervention Group) Participants in this arm will undergo standard surgical treatment for jaw cysts (enucleation with curettage) followed by adjunctive low-intensity pulsed ultrasound (LIPUS) therapy. Starting on the third postoperative day, LIPUS will be delivered using the OSTEOTRON IV device (Japan) at a frequency of 1.5 MHz and an intensity of 30 mW/cm². Each treatment session will last 20 minutes, applied once daily for 10 consecutive days. A trained nurse will administer the therapy under standardized conditions, with patients in a supine position and a coupling gel applied to the skin overlying the surgical site.
  The LIPUS intervention is expected to stimulate bone regeneration, reduce postoperative pain and numbness, and improve patients' overall recovery and quality of life compared with surgery alone.
  Interventions: Device: Low-Intensity Pulsed Ultrasound
- Sham-LIPUS therapy (Sham Comparator): Patients in the sham-LIPUS group underwent the same surgical procedure and received the same postoperative care as the ultrasound group. Beginning on the third day after surgery, they attended 10 daily sessions of sham treatment, each lasting 20 minutes. During these sessions, the same OSTEOTRON IV device was used, but it was deactivated so that no ultrasound waves were delivered. The device was applied to the skin over the cyst site with coupling gel in a controlled environment, mimicking the active treatment procedure.
  This design ensured that patients experienced the same setup, duration, and sensations of treatment without receiving the therapeutic ultrasound, thereby maintaining blinding and allowing a direct comparison with the active LIPUS group.
  Interventions: Device: Low-Intensity Pulsed Ultrasound

INTERVENTIONS:
Device: Low-Intensity Pulsed Ultrasound — The LIPUS therapy protocol was administered by a trained nurse following standardized procedures. Starting on the third day post-enucleation, patients in the ultrasound group underwent LIPUS therapy using the OSTEOTRON IV device (Japan), set at a frequency of 1.5 MHz and an intensity of 30 mW/cm², with 20-minute sessions for 10 consecutive days (Fig. 1). Treatments were conducted in a temperature-controlled environment, with patients positioned supine. Prior to each session, the skin over the cyst site was cleansed and coated with ultrasound transmission gel (Hinuo, Qingdao, China).

SUMMARY:
This study tested whether low-intensity pulsed ultrasound (LIPUS) could help patients recover better after surgery to remove jaw cysts.

A total of 29 patients with 33 jaw cysts were included. After surgery, they were randomly assigned to two groups:

Ultrasound group (17 patients, 18 cysts): received daily LIPUS therapy for 10 days.

Control group (12 patients, 15 cysts): received the same care but with a sham (inactive) device.

The study was triple-blinded, meaning that the patients, the surgeon, and the evaluators did not know who was receiving real or sham treatment.

Researchers measured recovery in several ways:

Patient reports: pain, numbness, anxiety/depression, and oral health-related quality of life.

Clinician monitoring: checked for any side effects (like infection or burns). Imaging tests (CBCT scans): tracked how well bone healed by measuring changes in cyst cavity size (volume reduction) and new bone density.

All patients had the same type of surgery, performed by the same surgeon, and all provided written informed consent. The study followed international ethics and trial registration standards.

DETAILED DESCRIPTION:
This clinical trial will explore whether a special type of ultrasound treatment, called low-intensity pulsed ultrasound (LIPUS), can improve recovery after surgery to remove cysts in the jaw. Jaw cysts are fluid-filled sacs that can weaken the jawbone, cause swelling, and sometimes lead to pain or numbness. The standard treatment is surgical removal of the cyst, but healing can take a long time, and patients may continue to experience discomfort or reduced quality of life.

To investigate a possible solution, researchers will enroll 29 patients with a total of 33 jaw cysts. After their cysts are surgically removed, patients will be randomly divided into two groups:

The ultrasound group will receive 10 days of daily LIPUS therapy, beginning three days after surgery.

The control group will receive the same routine care but with a sham (inactive) device that looks and feels the same, so patients will not know if they are receiving real ultrasound.

The study will use a triple-blind design, meaning that the patients, the surgeon, and the evaluators will not know which group each patient is in. This ensures that the results are as reliable and unbiased as possible.

Recovery will be evaluated in several ways:

Patient experiences: Participants will report on their pain levels, numbness, anxiety, depression, and overall quality of life using standard questionnaires.

Medical monitoring: Doctors will check for side effects such as infection, skin irritation, or other complications.

Advanced imaging: Cone-beam CT (CBCT) scans will measure how much the cyst cavity shrinks and how well new bone forms. The scans will also be used to track bone density over time, which shows how strong and healthy the healing bone becomes.

All surgeries will be performed by the same experienced surgeon to ensure consistency. The study will follow strict international research standards, including ethics approval and clinical trial registration. All participants will be fully informed about the study and will provide written consent before joining.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years.
* having undergone cyst enucleation with curettage.
* postoperative histopathological confirmation of a jaw cyst.
* willingness to complete 10 days of standardized LIPUS therapy

Exclusion Criteria:

* severe psychiatric disorders impairing compliance.
* acute infection.
* presence of a cardiac pacemaker.
* osteoporosis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2025-10-22 (Estimated); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
cyst cavity volume reduction | Time Frame: Measured from baseline (before cyst enucleation) to 3 months and 6 months post-treatment.
  The primary outcome measure of this trial will be cyst cavity volume reduction, assessed using cone-beam computed tomography (CBCT). Volumetric measurements of the cystic cavity (preoperative) and the residual cavity (at 3 and 6 months post-treatment) will be performed with Mimics 21.0 software (Materialise, Belgium).
Bone Density (CBCT, Relative Hounsfield Units). | Measured at baseline (pre-surgery), 3 months, and 6 months post-treatment.
  CBCT scans will quantify the mineral density of newly formed bone in the cyst site. The density will be expressed as relative Hounsfield Units (HU), using the nearest tooth's dentine as an internal reference. A relative HU value approaching 1 indicates higher bone mineralization, reflecting better bone regeneration after surgery with or without LIPUS therapy.

SECONDARY OUTCOMES:
Pain Intensity (VAS, 0-10) and Numbness Intensity (scale, 0-10) | Recorded before LIPUS/sham therapy, on Day 5, Day 10, 3 months, and 6 months post-treatment.
  Participants will rate the severity of pain at the surgical site, reflecting their comfort and recovery progress.
Oral Health-Related Quality of Life (OHIP-14, 0-56) | Pre-treatment, Day 10, 3 months, 6 months post-treatment.
  Measures functional limitations, pain/discomfort, and psychosocial impact related to oral health.

CONTACTS AND LOCATIONS:
Overall Officials: long jie, PhD, Principal Investigator — Sichuan University

IPD SHARING:
Plan to Share IPD: Undecided
The research team may reconsider data sharing in the future once appropriate safeguards and approvals are established."

REFERENCES:
- [Result] Wei Y, Guo Y: Clinical applications of low-intensity pulsed ultrasound and its underlying mechanisms in dentistry. Applied Sciences 2022, 12(23):11898.
- [Result] Gopalan A, Panneerselvam E, Doss GT, Ponvel K, Raja Vb K. Evaluation of Efficacy of Low Intensity Pulsed Ultrasound in Facilitating Mandibular Fracture Healing-A Blinded Randomized Controlled Clinical Trial. J Oral Maxillofac Surg. 2020 Jun;78(6):997.e1-997.e7. doi: 10.1016/j.joms.2020.01.036. Epub 2020 Feb 8. PMID 32145206
- [Result] Busse JW, Bhandari M, Kulkarni AV, Tunks E. The effect of low-intensity pulsed ultrasound therapy on time to fracture healing: a meta-analysis. CMAJ. 2002 Feb 19;166(4):437-41. PMID 11873920
- [Result] Lou S, Lv H, Li Z, Zhang L, Tang P. The effects of low-intensity pulsed ultrasound on fresh fracture: A meta-analysis. Medicine (Baltimore). 2017 Sep;96(39):e8181. doi: 10.1097/MD.0000000000008181. PMID 28953676